CLINICAL TRIAL: NCT04932694
Title: Optimizing Function Outcomes After Bariatric Surgery With Core Stabilization Training: A Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Batterjee Medical College (Other); Taif University (Other)
Responsible Party: Principal Investigator, Olfat Ibrahim Ali, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Bariatric Surgery
Record Dates: First submitted 2021-06-12; First posted 2021-06-21 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Bariatric Surgery; Surgery
Keywords: Bariatric surgery; Core training; Stabilization exercises
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Core stabilization exercises will be conducted for 8 weeks, 3 sessions per day at home, and exercises will be supervised remotly.
  Interventions: Other: Core stabilization training
- Control group (No Intervention): No exercise will be given to the participants in the control group

INTERVENTIONS:
Other: Core stabilization training — Exercise training will be given to the participants in the study group in the form of core training exercises for 8 weeks.
  Other Names: Exercises
  Arms: Study group

SUMMARY:
Bariatric surgery has been reported to be the most effective treatment option for losing and maintaining body weight and improving comorbidities and mortality associated with morbid obesity. Nevertheless, even though physical activity is recommended to optimize bariatric surgery results. Very little is known, about whether engaging in an exercise program after surgery can provide additional improvement in health outcomes. While to date there are relatively few researches studied the effect of exercise in patients who have undergone bariatric surgery.

DETAILED DESCRIPTION:
This study will investigate the effect of core stabilization exercise on patients who underwent bariatric suergery.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female
* age ranged from 18-25 years old,
* at least 6 months after BS

Exclusion Criteria:

* Patients with nerve root compression
* spine disorders
* spinal fracture
* previous spinal surgery
* pregnancy
* lower limb injury
* Any contraindication to the exercise therapy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
Core endurance tests | 2 months
  These tests consisted of four positions and calculated the time spent during the test.
Flexor extensor isokinetic torque | 2 months
  These tests consist of flexor and extensor isokinetic torque assessment.

SECONDARY OUTCOMES:
Balance assessment | 2 months
  assess the body balance using balance biodex system
6 min walking test | 2 months
  Assess aerobic capacity and endurance by measuring the distance covered in 6 minutes
Function Assessment | 2 months
  Assess function disability using Oswestry disability index questionnaire.
Trunk sense of position | 2 months
  Assess position sense of the trunk

CONTACTS AND LOCATIONS:
Overall Officials: Olfat I Ali, PhD, Principal Investigator — Cairo University
Locations (2):
- Olfat Ibrahim Ali, Giza, Dokki, Egypt
- Olfat Ibrahim Ali, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
Participants data will not be shared.